CLINICAL TRIAL: NCT00909701
Title: Investigating the Metabolic Response Following Intake of 2 Metabolic Preconditioning Drinks: a Randomized Double-blind Crossover Healthy Volunteer Study
Brief Title: Metabolic Response Following Intake of 2 Metabolic Preconditioning Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Enhanced Recovery After Surgery Group (part of ESPEN) (Unknown)
Responsible Party: Mr. Paul Cartledge, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B/12/2008
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Starvation
Keywords: Dietary supplement; healthy volunteers; Anaesthesia for surgery
MeSH Terms: conditions — Starvation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): PreOP Booster (Fresenius Kabi, Bad Homburg, Germany)
  Interventions: Dietary Supplement: PreOP Booster
- Comparator (Active Comparator): PreOP (Nutricia Clinical Care, Trowbridge, UK)
  Interventions: Dietary Supplement: PreOP (Nutricia Clinical Care, Trowbridge, UK)

INTERVENTIONS:
Dietary Supplement: PreOP Booster — 1 serving of 400 ml per study arm
  Arms: Test
Dietary Supplement: PreOP (Nutricia Clinical Care, Trowbridge, UK) — 1 serving of 400 ml per study arm
  Arms: Comparator

SUMMARY:
Surgical patients are usually starved for 8 to 12 hours before operation in order to reduce the chances of vomiting and other complications during the anaesthetic. Recent studies have suggested that this period of starvation might be harmful as it 'weakens' or 'stresses' the body before the operation. To avoid these harmful effects of starvation, patients are now given carbohydrate drinks (sugar-containing drinks that provide energy for the body) up to 2 hours before the operation. These drinks have been shown to make patients feel better, reduce sickness after the anesthetic/surgery and result in quicker recovery from operation. But the ways in which the sugar drinks have these beneficial effects on the body are unknown. The optimum time of giving these drinks to patients before operation is also unknown. This study will investigate the hormone responses of the body, following intake of 2 different carbohydrate drinks, in order to determine the optimum time of intake of these drinks in order to obtain the maximum benefits for the body.

ELIGIBILITY:
Inclusion Criteria:

* healthy male Caucasian volunteers aged 18-40 years,
* BMI of 20-25 kg/m2,
* able to give voluntary written informed consent to participate in the study, - able to understand the requirements of the study, including anonymous publications, AND
* agree to co-operate with the study procedure.

Exclusion Criteria:

* any history of acute or chronic illness, smoking, regular medication or substance abuse, OR
* have taken part in any other clinical study within the previous 3 months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
changes in plasma insulin and glucose levels | For 6 hours after intake of drink (blood samples will be taken at 20 min intervals for a total of 6 hours)

SECONDARY OUTCOMES:
Changes in plasma glucagon, non-esterified fatty acids and beta-hydroxybutyrate concentrations | For 6 hours after intake of drink (blood samples will be taken at 20 min intervals for a total of 6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Lobo, FRCS, Study Chair — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre Biomedical Research Unit, Nottingham, Nottinghamshire, United Kingdom